CLINICAL TRIAL: NCT01028638
Title: 89Zr-bevacizumab PET Imaging in Patients With Renal Cell Carcinoma Treated With Everolimus; a Pilot Study
Brief Title: Vascular Endothelial Growth Factor (VEGF) Imaging Before and During Everolimus Treatment for Renal Cell Carcinoma
Acronym: Everolimage
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: NL28799.042.09; METc2009.236
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: VEGF imaging; everolimus; renal cell carcinoma; PET; bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, white blood cells, plasma, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Renal Cancer: Renal Cancer patients treated with everolimus
  Interventions: Other: 89Zr-bevacizumab PET scan

INTERVENTIONS:
Other: 89Zr-bevacizumab PET scan — A tracer dose of 89Zr-bevacizumab (37 MBq, 5 mg protein dose) is given intravenously at day -3, day 11 and day 39.
  PET scans are made on day 1, day 15 and day 43.
  Other Names: VEGF imaging

SUMMARY:
Everolimus indirectly inhibits angiogenesis by reducing VEGF production. VEGF can be non-invasively visualized and quantified with serial 89Zr-bevacizumab PET imaging in patients.

The investigators hypothesize that a decline in VEGF early during everolimus treatment in patients with metastatic renal cell carcinoma predicts treatment efficacy.

89Zr-bevacizumab PET scans will be performed at baseline, after 2 and 6 weeks of everolimus treatment in 14 adult patients with metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
Background of the study

The majority of renal cell carcinomas (RCC) is characterized by profound angiogenesis because of inactivation of the Von Hippel Lindau gene. Angiogenesis inhibitors are established first line treatment options in the metastatic setting. Patients with progressive disease during or after treatment with angiogenesis inhibitors can benefit from treatment with everolimus, an oral mTOR inhibitor that resulted in doubling of progression free survival in a phase III study. Currently it is not possible to predict which patient will benefit from treatment with mTOR inhibitors. A predictive biomarker for efficacy of mTOR inhibitors is urgently needed as it may spare the patients unnecessary side effects, safes costs for the society as mTOR inhibitors are very expensive agents, and may speed up research on new drugs, drug combinations and drug dosing. One of the actions of mTOR inhibitors is blockage of production of vascular endothelial growth factor (VEGF), and this is thought to be the primary mechanism that is responsible for antitumor activity in RCC. The investigators hypothesize that non-invasive measurement of VEGF in the tumour and its surroundings by 89Zr-bevacizumab PET imaging before and shortly after start of everolimus is a good readout of efficacy of everolimus in patients with RCC.

Objective of the study

The primary objective of the study is to evaluate the feasibility of 89Zr-bevacizumab PET imaging as a biomarker before and during treatment with everolimus in patients with metastatic RCC. 89Zr-bevacizumab PET imaging will be regarded a promising biomarker if uptake changes after institution of treatment.

Study design

This is a pilot study for evaluation of 89Zr-bevacizumab PET imaging as a biomarker during treatment with everolimus in patients with mRCC.

89Zr-bevacizumab PET imaging will be performed before start of treatment and after 2 and 6 weeks of treatment.

Study population

14 patients who will start treatment with everolimus for metastatic RCC will be included in this study.

Primary study parameters

The primary endpoint is change in 89Zr-bevacizumab uptake in tumor lesions between the baseline scan and the scan during treatment.

Secondary study parameters The secondary endpoint is progressive disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, after 3 months of treatment. Progression is defined as the appearance of new disease or an increase of 20% in the sum of the longest diameters of the target lesions.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness

Patients will be intravenously injected at 3 time points with 37MBq resulting in a cumulative radiation dose of 54 mSv. According to ICRP 62 this radiation dose falls in category III (moderate risk).

Life expectancy of the patients is limited because of their incurable renal cell carcinoma, making the risk of development of a secondary malignancy clinically likely not relevant.

Patients have to pay 3 extra visits to the hospital for tracer injection. PET scans will be performed on regular visit days. Blood samples for biomarkers will be drawn during routine blood investigations.

There is no direct benefit for the patients in this study. If 89Zr-bevacizumab PET imaging however is a predictive biomarker for angiogenesis inhibitors, many patients can be spared unnecessary side effects and society can be spared costs of futile treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* metastatic renal cell cancer
* Intention to start treatment with everolimus
* WHO performance score ≤ 2
* measurable disease with x-ray or CT scan, at least one site of disease must be unidimensionally measurable as follows: X-ray > 20 mm Spiral CT scan > 10 mm Non-spiral CT scan > 20 mm
* ≥ 18 years
* not pregnant or nursing
* women of childbearing potential must use effective contraception
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* before patient randomization, written informed consent must be given according to GCP, and local regulations

Exclusion Criteria:

* formulated as "not" or "absence of" under inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic renal cell carcinoma who will start treatment with everolimus.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in 89Zr-bevacizumab uptake in tumor lesions between the baseline scan and the scan during treatment | Baseline, 2 weeks and 6 weeks

SECONDARY OUTCOMES:
Progressive disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, after 3 months of treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sjoukje Oosting, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] van Es SC, Brouwers AH, Mahesh SVK, Leliveld-Kors AM, de Jong IJ, Lub-de Hooge MN, de Vries EGE, Gietema JA, Oosting SF. 89Zr-Bevacizumab PET: Potential Early Indicator of Everolimus Efficacy in Patients with Metastatic Renal Cell Carcinoma. J Nucl Med. 2017 Jun;58(6):905-910. doi: 10.2967/jnumed.116.183475. Epub 2017 Jan 12. PMID 28082434